CLINICAL TRIAL: NCT05674045
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Dose-exploration Phase II Trial to Evaluate the Efficacy and Safety of EG017 Tablets in Postmenopausal Women With Stress Urinary Incontinence
Brief Title: A Phase 2, Randomized, Placebo-controlled, Double-blind Study of EG017 in Female Patients With Stress Urinary Incontinence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GenSci1002021II
Record Dates: First submitted 2022-12-30; First posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-10

CONDITIONS: Stress Urinary Incontinence
Keywords: stress urinary incontinence; Selective Androgen Receptor Modulator (SARM)
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- EG017 3mg (Experimental)
  Interventions: Drug: EG017 3mg
- EG017 6mg (Experimental)
  Interventions: Drug: EG017 6mg
- EG017 9mg (Experimental)
  Interventions: Drug: EG017 3mg; Drug: EG017 6mg
- Placebo Comparator: matching placebo (Placebo Comparator)
  Interventions: Drug: EG017 3mg; Drug: EG017 6mg

INTERVENTIONS:
Drug: EG017 3mg — EG017 3mg/day Oral administration for 12 weeks, once daily
  Arms: EG017 3mg; EG017 9mg; Placebo Comparator: matching placebo
Drug: EG017 6mg — EG017 6mg/day Oral administration for 12 weeks, once daily
  Arms: EG017 6mg; EG017 9mg; Placebo Comparator: matching placebo

SUMMARY:
The purpose of this study is to determine whether EG017 is safe and effective in the treatment of stress urinary incontinence in postmenopausal women.

DETAILED DESCRIPTION:
The main purpose of this study is to assess the efficacy of EG017 in female patients with stress urinary incontinence (SUI) compared with placebo as measured by the percent change in the urinary incontinence volume measured in a 1-hour pad test from baseline at week 12.

ELIGIBILITY:
Inclusion Criteria:

SUI symptoms of at least 6 months duration Urinary incontinence in the 1-hour pad test weight≥5g and<30 g Moderate to severe urinary incontinence evaluated by ICIQ-SF

Exclusion Criteria:

Patient has been diagnosed with mixed urinary incontinence (MUI) that is predominantly UUI Patient is considered to have SUI that would not be expected to improve unless treated with surgical therapy Patient had a history of surgical treatment for urinary incontinence (Trans-obturator tape surgery, Tension-free vaginal tape surgery, etc.) Patient has stage II or more of Pelvic Organ Prolapse (POP), or had a history of POP repair surgery before prior to study entry Patient has a serious illness or medical condition

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2022-09-26 (Actual)

PRIMARY OUTCOMES:
the percent change in the urinary incontinence volume measured in a 1-hour pad test | Baseline, week 12

SECONDARY OUTCOMES:
The percent change in urinary incontinence volume measured in a 24-hour pad test | Baseline, week 12
The percent change in urinary incontinence volume measured in 1-hour and 24-hour pad test | Baseline, week 8 week20
The average urinary incontinence episode frequency per 24 hours | Baseline, week 8, week 12, week20
The change in the international Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) | Baseline, week 8, week 12,week20
The change in UDI-6 scores | Baseline, week 8, week 12,week20
The change in PISQ-6 scores | Baseline, week 8, week 12,week20
Incidence of adverse events and side effects | Up to 20 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- People's Hospital of Peking University, Beijing, Beijing Municipality, China